CLINICAL TRIAL: NCT06833411
Title: Treatment for Giant Cell Arteritis With Tocilizumab and 8 as Compared to 26 Weeks of Prednisone: a Randomized, Multicenter, Adaptive, Blinded, Phase III Study
Brief Title: Treatment for Giant Cell Arteritis With Tocilizumab and 8 as Compared to 26 Weeks of Prednisone
Acronym: GISCO
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GISCO
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Giant Cell Arteritis (GCA)
Keywords: Tocilizumab; Glucocorticoid; Prednisone; Giant cell arteritis
MeSH Terms: conditions — Giant Cell Arteritis | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 26 weeks glucocorticoid (Active Comparator): 26 weeks glucocorticoid taper
  Interventions: Drug: Prednisone
- 8 weeks glucocorticoid (Experimental): 8 weeks glucocorticoid taper
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — Participant randomization to receive shortened (8 weeks) glucocorticoid taper upon initiation of a glucocorticoid-sparing agent.
  Arms: 8 weeks glucocorticoid
Drug: Prednisone — Participant randomization to receive standard (26 weeks) glucocorticoid taper upon initiation of a glucocorticoid-sparing agent.
  Arms: 26 weeks glucocorticoid

SUMMARY:
The GISCO study plans to determine whether 8-week therapy is just as effective as 26-week cortisone therapy for treating giant cell arteritis

* with tocilizumab,
* while using less cortisone.

DETAILED DESCRIPTION:
The aim of this randomized clinical trial investigates whether 1) a shortened GC 8-week regimen is as effective as the current 26-week regimen and 2) associated with less GC exposure when introducing a GC-sparing agent in the treatment of GCA.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with giant cell arteritis
* Start of tocilizumab treatment at baseline as part of routine clinical practice
* Receive ≥ 20 mg/day prednisone (or equivalent) at baseline
* Written informed consent

Exclusion Criteria:

* Treated with any investigational drug of chemical or biologic nature within a minimum of 30 days or 5 half-lives (whichever is longer) prior to the first dose of tocilizumab.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2032-08 (Estimated)

PRIMARY OUTCOMES:
Absence of a major relapse from randomization to 52 weeks | 52 weeks
  Composite endpoint. Pairwise comparisons of each patient from the control arm with each patient of the experimental arm.
Cumulative glucocorticoid exposure from randomization to 52 weeks | 52 weeks
  Composite endpoint. Pairwise comparisons of each patient from the control arm with each patient of the experimental arm.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Christ, Dr. med., Principal Investigator — Department of Rheumatology and Immunology, Inselspital, University of Bern, Bern, Switzerland
Locations (1):
- Department of Rheumatology and Immunology, Inselspital, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No